CLINICAL TRIAL: NCT06261788
Title: Efficacy and Safety of the Sync-AV II Temporary Cardiac Pacing Catheter (EASY II Trial)
Brief Title: Efficacy and Safety of the Sync-AV II Temporary Cardiac Pacing Catheter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swift Sync, Inc. (Industry)
Collaborators: Regulatory and Quality Solutions (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: EASY II Trial
Record Dates: First submitted 2024-01-31; First posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Heart Block; Valve Heart Disease
MeSH Terms: conditions — Heart Block; Heart Valve Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Temporary pacing — Transvenous temporary cardiac pacing - right internal jugular insertion

SUMMARY:
This is a prospective, single-center, non-randomized open label study. The objective of this study is to evaluate the efficacy and safety of the Sync-AV II Temporary Cardiac Pacing Catheter in subjects whose elective surgical or interventional procedure require temporary pacing support.

DETAILED DESCRIPTION:
The study will enroll up to 31 subjects at one investigational site with at least 3 implanters.

The subjects enrolled will be followed 7 days after the Sync-AV II Temporary Cardiac Pacing Catheter is removed. A safety call or clinic visit at 7 days post discharge will be performed.

Only subjects who meet the inclusion/exclusion criteria and provide informed consent will be eligible to receive the treatment and participate in the study. potential subjects who have a surgical or interventional procedure that will require temporary cardiac pacing support for at least 24 hours per investigator's medical judgement.

The elective surgical or interventional procedure is to be performed per institutional standard of care. Other concomitant therapy (medication and non-medication therapies) may be used during the study for the treatment or prevention of disease or to maintain good health.

Study Procedure standard of care technique to access the right jugular vein. Thru an introducer the Sync-AV II Temporary Cardiac Pacing Catheter is inserted Confirm and document the leads location as a baseline reference.

Acute Pacing Evaluation Acute pacing threshold evaluation will be performed immediate after leads deployed and at the end of the concomitant procedure.

Pacing Support During Concomitant Procedure Pacing setting to support for subject's medical need during concomitant procedure is per investigator's discretion.

Pacing Support During Hospital Stay Pacing setting to support for subject's medical need during hospital stay is per investigator's discretion.

Pacing Evaluation prior to Lead Removal Pacing lead evaluation will be performed immediately prior to the pacing catheter removal. The evaluation protocol will be the same as the lead evaluation at 24 hours post implant.

End of Study Subjects will exit the study after 7 days follow-up post procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is undergoing a surgical or an interventional procedure requiring temporary cardiac pacing to support for at least 24 hours per investigator's medical judgement.
2. Subject is at least 18 years of age.
3. Subject or legal representative provides written informed consent to the study.

Exclusion Criteria:

1. Subject has a co-exist temporary pacing or an implanted active permanent pacemaker or a cardiac defibrillator.
2. Subject on cardiogenic shock.
3. Subject is currently in atrial fibrillation.
4. Subject is pregnant or breastfeeding.
5. Subject had a stroke within 6 months prior to enrollment.
6. Subject has renal insufficiency with creatinine >2 mg/dl.
7. Subject with known bleeding diathesis.
8. Subject with a history of deep vein thrombosis or pulmonary embolization within 6 months.
9. Subject with known tricuspid valve disease that may impede catheter advance to and withdrawn from right ventricle.
10. Subject with known intracardiac thrombus or vegetation on echocardiography
11. Subject with significant neck abnormalities such that placement of a right and/or left internal jugular vein line would be difficult.
12. Subject has an active systemic infection or local infection at or around the insertion site.
13. Subject is involved in another clinical study that could influence the safety or outcome measures of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-09-13 (Actual); Study Completion 2023-09-26 (Actual)

PRIMARY OUTCOMES:
With a commercially available pacing box and/or analyzer, measure the ventricular pacing threshold at 24 hours post implant of the investigational device (index procedure) | 24 hours post implant
  Number of participants with a mean ventricular pacing threshold of less than 2.1 volts, measured at 24 hours post index procedure.
Procedure related complications | through study completion, an average of 7 days
  Incidence of serious procedural related complications
  The procedure-related serious complication is defined as:
  * Device-related endocarditis
  * Clinically significant cardiac perforation
  * New pericardial effusions requiring intervention
  * Sustained ventricular or atrial arrhythmia
  * Cardiac tamponade
  * Bleeding requiring transfusion

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Intervenciones Endovasculares y Cirugia Cardiovascular, Asunción, Paraguay

IPD SHARING:
Plan to Share IPD: Undecided
will be determined by board of directors at a later time

REFERENCES:
- [Background] Tancredi RG, McCallister BD, Mankin HT. Temporary transvenous catheter-electrode pacing of the heart. Circulation. 1967 Oct;36(4):598-608. doi: 10.1161/01.cir.36.4.598. No abstract available. PMID 6041872
- [Background] Lamas GA, Orav EJ, Stambler BS, Ellenbogen KA, Sgarbossa EB, Huang SK, Marinchak RA, Estes NA 3rd, Mitchell GF, Lieberman EH, Mangione CM, Goldman L. Quality of life and clinical outcomes in elderly patients treated with ventricular pacing as compared with dual-chamber pacing. Pacemaker Selection in the Elderly Investigators. N Engl J Med. 1998 Apr 16;338(16):1097-104. doi: 10.1056/NEJM199804163381602. PMID 9545357
- [Background] Perez SA, Ebner B, Kall CMY, Mitrani R, de Marchena EJ. A novel temporary atrioventricular sequential pacing catheter-Characteristics and first-in-human application. J Card Surg. 2022 Oct;37(10):2991-2996. doi: 10.1111/jocs.16796. Epub 2022 Jul 28. PMID 35900290